CLINICAL TRIAL: NCT04809207
Title: The CF Wellness Program to Treat Fatigue
Brief Title: Acceptability, Feasibility and Preliminary Efficacy of CFWP to Treat Clinically Elevated Fatigue in Adults With CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: University of Washington (Other); Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00202780
Record Dates: First submitted 2021-03-18; First posted 2021-03-22 (Actual); Last update posted 2023-08-28 (Actual); Status verified 2023-08

CONDITIONS: Cystic Fibrosis; Fatigue
MeSH Terms: conditions — Cystic Fibrosis; Fatigue

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CF Wellness Program (Experimental): Participants will receive CF Wellness Program sessions.
  Interventions: Other: CF Wellness Program Sessions

INTERVENTIONS:
Other: CF Wellness Program Sessions — The intervention will last approximately 12 weeks. During this time, up to 9 coaching sessions will be delivered. Each will last approximately 45 - 60 minutes. Sessions will be delivered either by web-based video chat (e.g., Zoom) or by telephone. Sessions will cover content such as understanding the physiological, cognitive, affective, behavioral contributors to CF fatigue; understanding the role of physical activity/exercise and fatigue including the importance of balancing activity and rest periods; cognitive restructuring; addressing attention and interpretation processes contributing to fatigue; teaching techniques such as mindfulness meditation relaxation strategies, good sleep hygiene, and activity scheduling and behavioral activation; and engaging social support. Physical activity goals will be set each session. Participants will be encouraged to use the provided fitness tracker and to sync weekly prior the coaching session so that the results can inform session content.

SUMMARY:
This research is being done to learn more ways to treat non-respiratory symptoms in people with CF including fatigue, pain, mood, sleep problems and the use of a wellness program to treat them.

DETAILED DESCRIPTION:
This study aims to test the acceptability, feasibility and preliminary efficacy of a tailored intervention known as the CF Wellness Program (CFWP) to treat clinically elevated fatigue in adults with CF. This is a pre-post pilot intervention study of the CF-Wellness Program. This study is needed because fatigue negatively affects health-related quality of life and has been identified by those with CF as a symptom that needs to be addressed. The study will include approximately 50 participants and the intervention will last approximately 13 weeks.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Documentation of CF diagnosis in the medical record
* If prescribed a modulator (i.e., ivacaftor, lumacaftor/ivacaftor, tezacaftor/ivacaftor, & elexacaftor/tezacaftor/ivacaftor), have been on treatment for at least 4 weeks
* If prescribed medicine for psychiatric purpose, must be on treatment for at least 8 weeks
* Has access to a smartphone, tablet, and/or computer with access to internet
* Ability to understand/read/speak English
* Receives CF care at a participating CF Center
* Has a score of >4 on the Fatigue Severity Scale
* Not likely to start and/or change modulator treatments during the intervention period

Exclusion Criteria:

* Receiving antibiotic treatment for a pulmonary exacerbation 14 days prior to the screening or expected to start within 14 days after screening visit
* Is pregnant or less than 6 months postpartum (self-reported)
* Is currently participating in another interventional trial
* Contraindication for aerobic exercise (determined by treating physician including cardiovascular, pulmonary and/or musculoskeletal contraindications)
* Forced Expiratory Volume in 1 second percent predicted (FEV1pp) is <25% within last year
* Planning to transfer care to a non-participating CF Center before the post-intervention visit could be completed
* Will not be available to complete CF-Wellness sessions in a timely fashion (e.g., will be on extended travel)
* Has already participated in the CF Wellness Program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Proportion enrolled in the CF Wellness Program (CFWP) | Day 0
  Number of participants enrolled into the CFWP Intervention among those eligible.
Proportion of cognitive behavioral therapy (CBT) sessions completed | At approximately 13 weeks post intervention
  Mean of the number of completed cognitive behavioral therapy (CBT) sessions divided by the number of sessions expected per participant.
Proportion of weeks participant synced the fitness tracker watch to the Smartphone app | At approximately 13 weeks post intervention
  This will be measured as the mean of the number of syncs completed divided by the number expected per participant. The fitness tracker watch with smartphone app data will be used to assess the proportion of weeks participant synced the fitness tracker watch to the Smartphone app.

SECONDARY OUTCOMES:
Feasibility of the CF Wellness Program as assessed by the Intervention Feasibility and Acceptability questionnaire (iFAQ) for patients | At approximately 13 weeks post intervention
  This measure will be used to evaluate feasibility of the intervention program. This measure will include questions about the feasibility of the program and will be assessed by the 5 point Likert Scale: Strongly disagree, Disagree, Neither Agree or Disagree, Agree, Strongly Agree.
  The scores will be averaged within participants to get a total score and then across participants; a mean score of 4 on a 5-point scale will be considered high satisfaction with the intervention.
Acceptability of the CF Wellness Program as assessed by the Intervention Feasibility and Acceptability questionnaire (iFAQ) for patients | At approximately 13 weeks post intervention
  This measure will be used to evaluate acceptability of the intervention program. This measure will be assessed by the 5 point Likert Scale: Strongly disagree, Disagree, Neither Agree or Disagree, Agree, Strongly Agree.
  The scores will be averaged within participants to get a total score and then across participants; a mean score of 4 on a 5-point scale will be considered high satisfaction with the intervention.
Qualitative interview as assessed by thematic analysis | At approximately 13 weeks post intervention
  A semi-structured interview will be conducted by the research team about the CF Wellness Program overall, and each module specifically, to determine the participants' perceptions of the degree to which the intervention was engaging, feasible, acceptable and useful. Recommendations for improving the CF Wellness Program will be solicited. The interviews will be recorded and their transcripts will be thematically analyzed using Nvivo Statistical & Qualitative Data Analysis Software.
Mean change in fatigue as assessed by the Functional Assessment of Chronic Illness-Fatigue ( FACIT-F) Scale | Day 1 to approximately 13 weeks post intervention
  The Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) is a measure that assesses self-reported fatigue and its impact upon daily activities and function. The scale is a 13-item, easy to administer tool that measures an individual's level of fatigue during their usual daily activities over the past week. The level of fatigue is measured on a four point Likert scale (4 = not at all fatigued to 0 = very much fatigued). The total scores will be calculated and a score greater than 36 will indicate elevated fatigue.
Change in exercise capacity as assessed by the 1 Minute Sit to Stand Test (1MSTST) test and Fitness tracker watch | Day 1 to approximately 13 weeks post intervention
  The 1 Minute Sit to Stand Test (1MSTST) test is used to assess exercise capacity and leg muscle strength. The participants are required to rise from a chair with their arms across their chest as often as possible in one minute. The number of chair rises will be calculated.
  The heart rate recovery (HRR) will be captured after the 1MSTST. The participant will wear a fitness tracker that will track heart rate. The heart rate peak will be calculated as the mean heart rate The fitness tracker watch will also be used to track the average 7 day daily step count of the study participants in order to determine if there are changes in their activity levels throughout the intervention program.
Change self-reported sleep disturbance as assessed by the Pittsburgh Sleep Quality Index (PSQI) | Day 1 to approximately 13 weeks post intervention
  This measures sleep disturbance and usual sleep habits during the prior month. The Pittsburgh Sleep Quality Scale (PSQI) is a 19-item self-rated questionnaire for evaluating subjective sleep quality the previous month. The 19 questions are combined into 7 clinically-derived component scores, each weighted equally from 0-3. The 7 component scores are added to obtain a global score ranging from 0-21, with higher scores indicating worse sleep quality.
Change in self-reported pain as assessed by the Patient-Reported Outcome Measurement Information System (PROMIS) Pain Intensity scale | Day 1 to approximately 13 weeks post intervention
  The PROMIS(r) Pain Intensity instrument assesses how much a person hurts. The items in the Pain Intensity scale assess pain intensity utilizing a 7-day recall period (items include the phrase "the past 7 days") while the last item asks patient to rate their pain intensity "right now. Each item is rated on a scale ranging from 1 (had no pain) to 5 (very severe). A higher total score, indicates severe pain level.
Change in self-reported depression as assessed by the Patient Health Questionnaire Depression Scale (PHQ-8) | Day 1 to approximately 13 weeks post intervention
  This is a measure used for assessing and monitoring depression severity. The PHQ-8 is an eight item self-reported measure of depression. Each item is rated on a scale ranging from 0 (not at all) to 3 (nearly every day). Total score is the sum of individual eight items and ranges from 0 to 24, with higher scores indicating more severe depression symptoms. Total score of 0 to 5 indicates none to minimal depression, 6 to 10 indicates mild depression, 11 to 15 indicates moderate depression, 16 to 20 indicates moderately severe depression and 21 to 24 indicates severe depression.
Change in self-reported anxiety as assessed by the General Anxiety Disorder - 7 (GAD7) scale | Day 1 to approximately 13 weeks post intervention
  This is a measure initially developed to diagnose generalized anxiety disorder. The GAD-7 is a seven item, self-reported measurement of GAD severity. Each item is rated on a scale ranging from 0 (not at all) to 3 (nearly every day). Total score is the sum of individual seven items and ranges from 0 to 21, with higher scores indicating more severe anxiety symptoms. Total score of 0 to 5 indicates none to minimal anxiety, 6 to 10 indicates mild anxiety, 11 to 15 indicates moderate anxiety, 16 to 21 indicates severe anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Kristin Riekert, PhD, Principal Investigator — Johns Hopkins University; Chris Goss, MD, Principal Investigator — University of Washington
Locations (2):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No